CLINICAL TRIAL: NCT00563966
Title: The Stress Responses of Fetuses and Infants Whose Mothers Smoked During Pregnancy: Genes, Hormones and Psychological Modulators
Brief Title: The Stress Responses of Fetuses and Infants Whose Mothers Smoked During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: David Mankuta, Hadassah
Other Study IDs: smokingmothers-HMO-CTIL
Record Dates: First submitted 2007-11-25; First posted 2007-11-27 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2007-11

CONDITIONS: Effects of Smoking on Infant
Keywords: smoking pregnancy behaviour polymorphisms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples + salivery cortisol
Oversight: Data Monitoring Committee: No

SUMMARY:
It is generally understood that smoking during pregnancy has deleterious effects on the developing fetus, although research on smoking during pregnancy has been limited in focus, with most studies focused on birth weight of newborns and children's behavioral disturbances. However, little is known about the neurobiological underpinnings of nicotine-related developmental deficits and even less is known about genetic and environmental factors that may exacerbate the risk for such deficits in some children. In this study, we propose to examine the relation between antenatal exposure to nicotine and infants' stress-responses before and after birth (2-days, 6-months) and its moderation of by family-based stressors and genes related to nicotine metabolism and stress responsivity.

We hypothesize that the risk imposed on infants by antenatal exposure to nicotine is moderated by genotype that influences functioning of the HPA axis, metabolism of nicotine, and stress-levels and parenting that influence the development of neural substrates (HPA axis) and infants' capacity to cope with stress. There is a growing consensus that Gene x Environmental (G x E) interplay likely mediated by epigenetic effects constitute one of the central mechanism by which complex disorders develop. Our proposal offers an exceptional paradigm to explore the association between genes, environment, and G x E interactions on the neural and behavior response of children to stressful challenges.

DETAILED DESCRIPTION:
Detailed Description of the Proposed Research

Design overview. A large cohort of pregnant women will be recruited, and those who meet criteria will be divided into two groups according to their testimony regarding their smoking behavior and saliva cotinine screening, as in our previous studies. At 3-time points, the antenatal period, 2-days and 6-months of age; we will assess infants' responses to challenges using biochemical, behavioral, and subjective measures. The challenges selected are "proven" stressors and previous research has demonstrated their effectiveness in eliciting stress-reactions (e.g., increased cortisol). In parallel, we will obtain an obstetric history (from medical records), demographics, measure of symptomology, information on smoking and drinking habits, life stresses, and family cohesion at each time point, plus information about mothers' feelings/behavior and mothers' ratings of infants "regulatory" behavior after birth. The antenatal and neonatal sessions will be carried out in Hadassah Hospital and the 6-month session in the developmental laboratory at Hebrew University. Genetic material will be collected from parents and their infant at childbirth.

Recruitment Women smokers will be recruited will be recruited by nurses in well-baby clinics (where physicians do routine prenatal check-ups), gynecologists, midwives, and by advertisement. In addition, we will recruit women at the time of routine checks in Hadassah hospital (Nuchal translucency test) at 12 weeks, triple/quadra test blood testing at 16 weeks, early (14-16 weeks) and advanced (20-22 week) fetal anatomy scan, and glucose test at 24-28 weeks) (supervised by Dr. Mankuta). In all, we will recruit 150 women for the "smoking" group, using the following inclusion criteria: smokes at least 10 cigarettes a day (i.e., habitual smokers) no abuse of alcohol or drugs, no chronic physical disability, 22-35 years of age, living with partner, speaks English, Hebrew, or Russian, natural conception). A (second) group of 150 women who meet inclusion criteria (except smoking) and matched in age, education, gender of infant, and parity to the "smokers" will serve as controls. At recruitment and each time-point, mothers (and their spouses) who agree to participate in the research protocol will be interviewed for smoking habits (Fagerstrom Tolerance Questionnaire, FTQ) as detailed in our previous studies on smoking. At recruitment, women will be explicitly told that we are not encouraging smoking and will provide resources if, at any time, during the study, they want to stop smoking.

Antenatal period (Dr. David Mankuta)

The prenatal session will be carried out at 34-36 weeks of gestation (by last menstrual period and confirmed by early ultrasound) and will consist of 3 phases: (1) waiting room- in which mothers receive instructions, (2) ultrasound- to evaluate limb movement before and after vibroacoustic stimulation (VAS), as well as measures of fetuses' well-being (cardiotocograph test, biophysical profile), and (3) post exam- administration of questionnaires.

Limb movement. Measures of fetal limb movement are good reflections of infant state, are stable from late gestation out to 4-weeks postnatal age 80 , are affected by antenatal stress 81, and forecast infants' state regulation 2 weeks after birth. Ultrasound (ATL 3500 and 5000) will be used to visualize and film the fetus for offline coding of limb movements. To begin testing, infant must be in state 1F, characterized by minimal fetal movement for 2 minutes. When this criterion is met, baseline the VAS (Fetal Acoustic Corometrics Stimulator Model 146; ≈75 HZ, ≈82 db) will be presented for 5 s. Fetal movements will be videotaped with the recorder built into the scanner. During off-line time-event coding, each limb movement will be counted. From these raw counts, we will average the number of movements observed in 10 s intervals during the 1 min prior to (baseline) and during the 5 min after stimulation. Reactivity will be derived by calculating the difference between the mean baseline count and the mean count recorded during the 5 s of stimulation. Regulation will be calculated as (1) the slope of the counts across the post stimulation period (5 minutes), and (2) the difference between the mean baseline count and the mean count of last three 10 second epochs. for first time point. Previous studies have shown limb-counts to be stable (24-36 weeks), reliable, and sensitive to maternal stress.

Questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Smokes at least 10 cigarettes a day
* No abuse of alcohol or drugs
* No chronic physical disability
* 22-35 years of age
* Living with partner
* Speaks English, Hebrew, or Russian
* Natural conception

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who smoked during pregnancy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ebstein Richard, MD PhD, Study Chair — Hebrew University Jerusalem Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel